CLINICAL TRIAL: NCT07290010
Title: A Clinical Trial to Explore the Efficacy and Safety of Iparomlimab and Tuvonralimab Injection Combined With Chemotherapy as the First-line Treatment for Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: The Efficacy and Safety of Iparomlimab and Tuvonralimab Injection Combined With Chemotherapy as the First-line Treatment for Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025KY012
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: immunotherapy; ESCC; PD-1/CTLA-4; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab combined with chemotherapy (Experimental): Patients were enrolled and received 6 cycles of Iparomlimab and Tuvonralimab combined with albumin-bound paclitaxel and cisplatin. Subsequently, maintenance treatment was carried out using Iparomlimab and Tuvonralimab ± albumin-bound paclitaxel until disease progression or the occurrence of unacceptable adverse events
  1. Iparomlimab and Tuvonralimab Injection: 5 mg/kg, d1, Q3W;
  2. Albumin-bound paclitaxel:100-150 mg/m², d1, d8, Q3W;
  3. Cisplatin: 75 mg/m², d1, Q3W;
  Interventions: Drug: Iparomlimab and Tuvonralimab combined with chemotherapy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab combined with chemotherapy — Patients were enrolled and received 6 cycles of Iparomlimab and Tuvonralimab combined with albumin-bound paclitaxel and cisplatin. Subsequently, maintenance treatment was carried out using Iparomlimab and Tuvonralimab ± albumin-bound paclitaxel until disease progression or the occurrence of unacceptable adverse events 1. Iparomlimab and Tuvonralimab Injection: 5 mg/kg, d1, Q3W; 2. Albumin-bound paclitaxel:100-150 mg/m², d1, d8, Q3W; 3. Cisplatin: 75 mg/m², d1, Q3W;

SUMMARY:
This study is a single-arm clinical trial to evaluate the efficacy and safety of Iparomlimab and Tuvonralimab combined with chemotherapy in the first-line treatment of patients with recurrent or metastatic esophageal squamous cell carcinoma (ESCC). After screening and meeting the inclusion criteria, the patients were enrolled and received 6 cycles of Iparomlimab and Tuvonralimab combined with albumin-bound paclitaxel and cisplatin. Subsequently, maintenance treatment was carried out using Iparomlimab and Tuvonralimab ± albumin-bound paclitaxel until disease progression or the occurrence of unacceptable adverse events, with a total maximum treatment duration of 24 months.

The main objective of this study is to: 1. evaluate the ORR of Iparomlimab and Tuvonralimab combined with albumin-bound paclitaxel and cisplatin. 2. The secondary endpoints include PFS, DCR, DoR, OS and safety, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender not limited;
2. Unresectable, recurrent or advanced metastatic esophageal squamous cell carcinoma confirmed by histopathological examination (excluding adenosquamous carcinoma mixed type and other pathological types);
3. For patients who have previously received adjuvant/neoadjuvant chemotherapy/chemoradiotherapy, or radical concurrent chemoradiotherapy , the time from the last treatment to disease recurrence is more than 6 months;
4. ECOG 0-1;
5. According to RECIST v1.1, there is at least one measurable lesion;
6. Be capable of providing newly obtained or archived tissue samples for immunohistochemical analysis of PD-L1 expression;
7. The patient's organ functions are normal, with no serious abnormalities in blood, heart, lung, liver or kidney functions, and no immune deficiency diseases.
8. The patient has normal coagulation function and no active bleeding or thrombotic diseases.
9. Expected survival time ≥12 weeks;
10. Male subjects who are female of childbearing age or whose sexual partners are female of childbearing age must take effective contraceptive measures throughout the treatment period and for 6 months after the treatment period.
11. Voluntarily sign a written informed consent form and be able to comply with the visitation and related procedures stipulated in the plan

Exclusion Criteria:

1. Locally advanced esophageal cancer that can be potentially cured through radical surgical resection or radiotherapy;
2. Esophageal squamous cell carcinoma that is known to have complete obstruction under endoscopy and requires interventional treatment to relieve the obstruction;
3. There is a risk of perforation after stent implantation in the esophageal or tracheal cavity;
4. Has received systemic treatment for advanced or metastatic esophageal squamous cell carcinoma in the past;
5. Other malignant tumors diagnosed within 5 years prior to the first administration, except for effectively treated cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma and/or effectively resected cervical cancer and/or breast cancer in situ;
6. Severe infection occurs (CTCAE>grade 2), or active pulmonary inflammation;
7. Previous or current interstitial pneumonia, pneumoconiosis, drug-related pneumonia, or severe lung function impairment;
8. Patients with active tuberculosis infection;
9. Participate in another interventional clinical study simultaneously, unless participating in an observational (non-interventional) clinical study or being in the follow-up stage of an interventional study;
10. Patients with congenital or acquired immune deficiencies, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive hepatitis C antibody and HCV-RNA above the detection limit), or patients with co-infection of hepatitis B and hepatitis C;
11. There is a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
12. Having undergone major surgical operations (craniotomy, thoracotomy or laparotomy) within 4 weeks prior to the first dose of the study treatment or expecting to undergo major surgeries during the study treatment period;
13. It is known that there are symptomatic central nervous system metastases and/or cancerous meningitis (except for stable brain metastases that do not require steroid treatment);
14. It is known that there is an active autoimmune disease requiring symptomatic treatment or a history of the disease within the past 2 years (patients with vitiligo, psoriasis, alopecia or Graves' disease that do not require systemic treatment in the past 2 years, hypothyroidism who only need thyroid hormone replacement therapy, and type 1 diabetes who only need insulin replacement therapy can be enrolled).
15. Female patients who are pregnant or breastfeeding;
16. Any serious or uncontrolled systemic disease that researchers believe may increase the risk of participation in patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | 18months
  The objective response rate (ORR) evaluated by investigator based on RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival （PFS） | 24months
  The Progression-free survival (PFS) evaluated by investigator based on RECIST 1.1
Disease control rate (DCR) | 18months
  Disease control rate (DCR) evaluated by investigator based on RECIST 1.1
Duration of response (DoR) | 24months
  Duration of response (DoR) evaluated by investigator based on RECIST 1.1
Overall survival（OS） | 30months
  Overall survival（OS）
Adverse events（AEs） | 24months
  The incidence and severity of adverse events (AEs) : The incidence and severity of adverse events (AE) and serious adverse events (SAE) were determined based on the NCI-CTCAE v5.0 standard. Abnormal vital signs and laboratory tests, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No